CLINICAL TRIAL: NCT04083534
Title: Phase 1/2 FIH Study of REGN5459 (Anti-BCMA x Anti-CD3 Bispecific Antibody) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: First In Human (FIH) Study of REGN5459 in Adult Patients With Relapsed or Refractory Multiple Myeloma (MM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5459-ONC-1888; 2019-001108-39 (EudraCT Number)
Record Dates: First submitted 2019-08-29; First posted 2019-09-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- REGN5459 (Experimental): Cohorts of multiple REGN5459 dose levels
  Interventions: Drug: REGN5459

INTERVENTIONS:
Drug: REGN5459 — Administered by intravenous (IV) infusion

SUMMARY:
In the phase 1 portion of the study, the primary objectives are to assess the safety, tolerability, and dose-limiting toxicities (DLTs) and to determine a recommended phase 2 dose regimen (RP2DR) of REGN5459 as monotherapy in patients with relapsed or refractory multiple myeloma (MM) who have exhausted all therapeutic options that are expected to provide meaningful clinical benefit.

In the phase 2 portion of the study, the primary objective is to assess the preliminary anti-tumor activity of REGN5459 as measured by objective response rate (ORR).

In the phase 1 and phase 2 portion, the secondary objectives of the study are:

* To assess the preliminary anti-tumor activity of REGN5459 as measured by duration of response (DOR), progression-free survival (PFS), rate of minimal residual disease (MRD) negative status, and overall survival (OS)
* To evaluate the pharmacokinetic (PK) properties of REGN5459
* To characterize the immunogenicity of REGN5459
* To evaluate the effects of REGN5459 on patient-reported quality of life (QoL), symptoms, functioning and general health status

In the phase 1 portion of the study only, the secondary objective of the study is to assess the preliminary anti-tumor activity of REGN5459 as measured by ORR.

In the phase 2 portion of the study only, the secondary objective of the study is to evaluate the safety and tolerability of REGN5459.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Patients must have myeloma that is response-evaluable according to the 2016 International Myeloma Working Group (IMWG) response criteria
* Measurable disease is defined as 1 or more of the following:

  1. Serum M-protein ≥1 g/dL,
  2. Urine M-protein ≥200 mg/24-hour, and/or
  3. Free light chain (FLC) assay with involved FLC level ≥10 mg/dL with an abnormal serum FLC ratio
* A patient with Immunoglobulin A (IgA) myeloma but without measurable M-protein may be enrolled if quantitative IgA levels are ≥400 mg/dL and can be followed longitudinally
* A patient with non-secretory MM may be considered for enrollment after discussion with the sponsor that includes the feasibility of an individualized plan for response assessment
* Patients with MM who have exhausted all therapeutic options that are expected to provide meaningful clinical benefit, either through disease relapse, treatment refractory disease, or intolerance of the therapy, and including either:

  1. Progression on or after at least 3 lines of therapy, or intolerance of therapy, including a proteasome inhibitor, an Immunomodulatory imide drug (IMiD), and an anti-CD38 antibody, OR
  2. Progression on or after an anti-CD38 antibody and having disease that is "double refractory" to a proteasome inhibitor and an IMiD, or intolerance of therapy. The anti-CD38 antibody may have been administered alone or in combination with another agent such as a proteasome inhibitor. Refractory disease is defined as lack of response or relapse within 60 days of last treatment.
* Adequate hematologic function as measured by:

  1. Platelet count > 50 x 109/L. A patient may not have received a platelet transfusion within 7 days to meet this platelet eligibility requirement.
  2. ANC > 1.0 x 109/L. A patient may not have received granulocyte colony stimulating factor (G-CSF) within 2 days to meet this absolute neutrophil count eligibility requirement.
  3. Hemoglobin > 8.0 g/dL
* Adequate hepatic function, defined as:

  1. Total bilirubin ≤1.5 x ULN
  2. Transaminase (ALT, AST) ≤2.5 x ULN
  3. Alkaline phosphatase ≤2.5 x ULN
* Patients with Gilbert syndrome do not need to meet this total bilirubin requirement provided that the total bilirubin is unchanged from the baseline value.

  d. Serum creatinine clearance by Cockcroft-Gault >30 mL/min
* A patient with a creatinine clearance by Cockcroft-Gault who does not meet eligibility criteria may be considered for enrollment if a measured creatinine clearance (based on 24-hour urine collection or other reliable method) is >30 mL/min
* Life expectancy of at least 6 months

Key Exclusion Criteria:

* Patients with known MM brain lesions or meningeal involvement
* History of neurodegenerative condition or central nervous system (CNS) movement disorder, or patients with a history of seizure within 12 months before study enrollment are excluded
* Cardiac ejection fraction <40% by echocardiogram or multi-gated acquisition scan (MUGA)
* Prior treatment with any anti-BCMA antibody (including antibody-drug conjugate or bispecific antibody) or BCMA-directed CAR T therapy
* Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection; or other uncontrolled infection

  1. Patients with HIV who have controlled infection (undetectable viral load and CD4 count above 350 cells/microliter either spontaneously or on a stable antiviral regimen) are permitted.
  2. Patients with hepatitis B (Hepatitis B Surface Antigen Test positive [HepBsAg+]) who have controlled infection (serum HBV DNA polymerase chain reaction [PCR] that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted.
  3. Patients who are HCV antibody-positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by polymerase chain reaction (PCR) either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
* History of allogeneic stem cell transplantation at any time, or autologous stem cell transplantation within 12 weeks of the start of study treatment

NOTE: Other protocol defined Inclusion/Exclusion Criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) from the first dose through the end of the DLT observation period | Up to 35 Days
  Phase 1
Incidence and severity of treatment-emergent adverse events (TEAEs) during REGN5459 treatment period | Up to 12 Weeks After the Last Dose
  Phase 1
Incidence and severity of adverse events of special interest (AESI) with REGN5459 treatment period | Up to 12 Weeks After the Last Dose
  Phase 1
Objective response rate (ORR) as measured using the International Myeloma Working Group (IMWG) criteria | Up to Approximately 104 Weeks
  Phase 2

SECONDARY OUTCOMES:
Concentrations of REGN5459 in the serum over time | Up to 12 Weeks After the Last Dose
  Phase 1 and phase 2
Incidence over time of anti-drug antibodies (ADAs) to REGN5459 | Up to 12 Weeks After the Last Dose
  Phase 1 and phase 2
Duration of response (DOR) using the IMWG criteria | Up to Approximately 104 Weeks
  Phase 1 and phase 2
Progression-free survival (PFS) as measured using the IMWG criteria | Up to Approximately 104 Weeks
  Phase 1 and phase 2
Rate of minimal residual disease (MRD) negative status using the IMWG criteria | Up to Approximately 104 Weeks
  Phase 1 and phase 2
Overall survival (OS) | Up to Approximately 104 Weeks
  Phase 1 and phase 2
Patient-reported Quality of Life (QOL) per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Up to 12 Weeks After the Last Dose
  Phase 1 and phase 2
  The EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social) , symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Patient-reported QOL per EORTC Quality of Life Questionnaire-Multiple Myeloma module 20 (EORTC QLQ-MY20) | Up to 12 Weeks After the Last Dose
  Phase 1 and phase 2
  The EORTC QLQ-MY20 is a self-administered instrument to assess QoL in persons with MM. This 20-item questionnaire measures the following domains: symptom scales, including disease symptoms (6 items) and symptoms related to side effects of treatment (10 items); function scale and future perspective (3 items); and body image (1 item). A high score represents a high level of symptoms or problems.
Patient-reported QOL per EuroQoL-5 Dimension-3 Level Scale (EQ-5D-3L) | Up to 12 Weeks After the Last Dose
  Phase 1 and phase 2
  The EQ-5D-3L is a self-administered generic standardized health status measure, consisting of an EQ-5D descriptive system and an EQ visual analog scale. The EQ-5D-3L descriptive system assesses 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 3-level scale: no problems, some problems, and extreme problems. The EQ visual analog scale component is a vertical visual analog scale used by patients to rate their health.
Change in patient-reported global health status/QOL per EORTC QLQ-C30 | Baseline up to 12 Weeks After the Last Dose
  Phase 1 and phase 2
  The EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social) , symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Time to definitive deterioration in patient-reported global health status/QOL per EORTC QLQ-C30 | Up to 12 Weeks After the Last Dose
  Phase 1 and phase 2
  The EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social) , symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Change in patient-reported general health status per EQ-5D-3L | Baseline up to 12 Weeks After the Last Dose
  Phase 1 and phase 2
  The EQ-5D-3L is a self-administered generic standardized health status measure, consisting of an EQ-5D descriptive system and an EQ visual analog scale. The EQ-5D-3L descriptive system assesses 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 3-level scale: no problems, some problems, and extreme problems. The EQ visual analog scale component is a vertical visual analog scale used by patients to rate their health.
ORR as measured using the IMWG criteria | Up to Approximately 104 Weeks
  Phase 1 Only
Incidence and severity of TEAEs during REGN5459 treatment period | Up to 12 Weeks After the Last Dose
  Phase 2 Only
Incidence and severity of AESI during REGN5459 treatment period | Up to 12 Weeks After the Last Dose
  Phase 2 Only

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Investigator, Study Director — Regeneron Pharmaceuticals
Locations (7):
- United States (7):
  - Regeneron Study Site, Indianapolis, Indiana
  - Regeneron Study Site, Ann Arbor, Michigan
  - Regeneron Study Site, Rochester, Minnesota
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://errs.regeneron.com/external